CLINICAL TRIAL: NCT05792306
Title: A Novel Electrolyzed Water Spray Reduces Discomfort, Redness and Swelling of the Skin Surrounding the Wound Created by Skin Lasar Surgery: A Clinical Study
Brief Title: The Novel Electrolyzed Water Spray Treatment Discomfort, Redness and Swelling of the Skin Surrounding the Wound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jia19920107
Record Dates: First submitted 2023-02-27; First posted 2023-03-31 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-02

CONDITIONS: Skin Injury
Keywords: Electrolyzed water device; Hydroxyl radical; Tap water; Spray; Laser surgery wound; Discomfort of the skin; Redness of the skin

STUDY DESIGN:
Intervention Model Description: An open label, two arm clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The electrolyzed water spray group (Experimental): Study staff will use the novel electrolyzed water spray device and spray for approximately 2-4 minutes on the participant's diseased area until half a bottle (20-40ml) of water is used.
  Interventions: Device: The novel electrolyzed water spray
- Control group of water spray (Placebo Comparator): Study staff will use the saline and spray for approximately 2-4 minutes on the participant's diseased area until half a bottle (20-40ml) of water is used.
  Interventions: Device: The saline spray

INTERVENTIONS:
Device: The novel electrolyzed water spray — The researcher use electrolyzed water to treat the diseased area, two times a day, for 5 days. The trial consists of 5 study visits (day 1-day 5). The reduction in the disease area of discomfort, redness and swelling evaluation and adverse event assessments will be performed at each visit. Safety analysis will be assessed based on the reports of adverse events during the study.
  Arms: The electrolyzed water spray group
Device: The saline spray — The researcher use saline to treat the diseased area, two times a day, for 5 days. The trial consists of 5 study visits (day 1-day 5). The reduction in the disease area of discomfort, redness and swelling evaluation and adverse event assessments will be performed at each visit. Safety analysis will be assessed based on the reports of adverse events during the study.
  Arms: Control group of water spray

SUMMARY:
The purpose of this study is to test whether the reduction of the sense of discomfort and redness and swelling of the skin surrounding the wound of patients by use of the novel electrolyzed water spray will relieve the inflammation of the skin.

DETAILED DESCRIPTION:
In this study, water inculding tap water,pure water and salt water, and an apparatus for producing electrolyzed water (https://www.deposon.com.cn; https://www.deposon.com）were used to generate an electrolyzed water mist spray or spray. This instantly generated electrolyzed water mist spray or spray has oxidation-reduction potential (ORP) ≥1200mv,and contains non-specific total oxidation capacity which equals to 0.28±0.10ppm,0.06±0.04ppm and 3.92±0.39ppm of desolved ozone. This instantly generated electrolyzed water mist spray or spray does not release detectable ≥0.1mg/m3 of gaseous ozone. This instantly generated electrolyzed water mist spray or spray has pH 8.4±0.4 and releases negative air ion.The apparatus for producing electrolyzed water has a positive electrode which is covered by a conductive diamond material (Patent# CN215308550U). In this study, this novel electrolyzed water device and the water spray are used to treat wounds created by skin laser surgery.

ELIGIBILITY:
Inclusion Criteria:

* Mild discomfort, redness and swelling of the skin surrounding the wound created by skin laser surgery
* Patient > 18 years old.

Exclusion Criteria:

* Severe discomfort, redness and swelling of the skin surrounding the wound created by skin laser surgery.
* 80 years or older.
* Pregnant or breastfeeding women
* Systemically healthy individuals.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
The sense of discomfort scale made by the Numeric Pain Rating Scale (NPRS). | 1 hour
  This score is based on descriptions of the discomfort of the skin surrounding the wound that patients rate 0-10 to assess the condition of their skin. A higher score means a worse outcome. 0 means "no discomfort " and 10 means "the most discomfort ".

SECONDARY OUTCOMES:
A skin signs scale made by modifying the Numeric Pain Rating Scale (NPRS). | 3 hour
  The skin signs scale evaluations the signs of skin wound inflammation including redness and swelling of the skin immediately surrounding the wound. This score is based on descriptions of the redness and swelling of the skin surrounding the wound that patients rate 0-10 to assess the condition of their skin. A higher score means a worse outcome. 0 means "no redness and swelling of the skin surrounding the wound " and 10 means "the most redness and swelling surrounding the wound".

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: until publication of this clinical study and international patent granted